CLINICAL TRIAL: NCT01687309
Title: A Study to Investigate the Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of GSK2586184 Following a Single Doseof 800mg and Repeat Oral Tablet Doses of 800mg b.d and the Effect of Food and Gender on the Pharmacokinetics of oralGSK2586184 in Healthy Subjects
Brief Title: A Study to Investigate the Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of Single and Repeat Doses of GSK2586184 and the Effect of Food and Gender
Acronym: JAK116439
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 116439
Record Dates: First submitted 2012-05-10; First posted 2012-09-18 (Estimated); Last update posted 2018-05-25 (Actual); Status verified 2018-05

CONDITIONS: Systemic Lupus Erythematosus
MeSH Terms: conditions — Lupus Erythematosus, Systemic | interventions — GSK2586184; Single Person; Food

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- Cohort A fed session (Other): GSK2586184 800mg single dose with food
  Interventions: Other: GSK2586184 single dose taken with food
- Cohort A fasted session (Other): GSK2586184 single dose without food
  Interventions: Other: GSK2586184 single dose taken without food
- Cohort B active study medication (Active Comparator): GSK2586184 800mg single and twice daily dose for 13 days
  Interventions: Drug: GSK2586184 800mg single and repeat dose
- Cohort B placebo (Placebo Comparator): Placebo-to-match single and twice daily dose for 13 days
  Interventions: Drug: Placebo-to-match GSK2586184

INTERVENTIONS:
Drug: GSK2586184 800mg single and repeat dose — GSK2586184 800mg single dose and then twice daily dosing for 13 days
  Arms: Cohort B active study medication
Drug: Placebo-to-match GSK2586184 — Placebo-to-match GSK2586184
  Arms: Cohort B placebo
Other: GSK2586184 single dose taken with food — GSK2586184 single dose taken with FDA approved high fat, high calorie breakfast
  Arms: Cohort A fed session
Other: GSK2586184 single dose taken without food — GSK2586184 single dose taken in a fasted state
  Arms: Cohort A fasted session

SUMMARY:
A study to investigate the safety, tolerability, pharmacokinetics, and pharmacodynamics of single and repeat doses of 800 mg GSK2586184 in healthy subjects.

DETAILED DESCRIPTION:
This is a study in healthy volunteers to investigate the safety, tolerability, pharmacokinetics (the body's effect on the drug) and pharmacodynamics (the drug's effect on the body) of single and repeat doses of 800 mg GSK2586184. The effect of food and gender on pharmacokinetics will also be investigated following single dosing.

The study is made up of 2 groups of healthy subjects. The first group consists of 6 female subjects who will receive a single dose of 800mg GSK2586184 (study medication) during 2 seperate sessions. One session will involve the female subjects taking the study medication with food and the other session will involve study medication being taken without food. The safety and tolerability of the study medication in female subjects and the effect of food on the pharmacokinetics of the study medication will be investigated.

The second group will consist of 12 healthy male subjects participating in 2 sessions. 8 subjects will receive study medication and 4 will receive placebo (dummy medication) during the course of the study. Neither they or their study doctor will know which one they are given. Each male subject will receive a single dose of study medication or placebo followed by 13 days of twice daily dosing of study medication or placebo. Each dose will be taken with food.The single dose results from this group of subjects will be compared to the female group to investigate the effect of gender on pharmacokinetics. The safety and pharmacokinetics of repeat dosing will be investigated. The effect of repeat dosing on kidney function and the immune system will also be investigated.

The study will take place in the SGS Clinical Pharmacology Unit in Antwerp, Belgium. A pharmaceutical company, GlaxoSmithKline, is funding the study.

ELIGIBILITY:
Inclusion Criteria:

* Healthy as determined by a responsible and experienced physician, based on a medical evaluation including medical history, physical examination, laboratory tests and cardiac monitoring
* Cohort A: A female subject of non-childbearing potential defined as pre-menopausal females with a documented tubal ligation or hysterectomy; or postmenopausal defined as 12 months of spontaneous amenorrhea
* Cohort B: Male subjects with female partners of child-bearing potential must agree to contraception method mandated by protocol
* Cohort A: Subjects between 18 and 65 years of age inclusive, at the time of signing the informed consent
* Cohort B: Subjects between 18 and 50 years of age inclusive, at the time of signing the informed consent
* Normal creatinine clearance values at screening
* ALT, alkaline phosphatase and bilirubin ≤ 1.5xULN (isolated bilirubin >1.5xULN is acceptable if bilirubin is fractionated and direct bilirubin <35%)
* Single QTcF < 480 msec
* BMI within the range 18 - 30.0 kg/m2 (inclusive)
* Subjects must be non-smokers and must not use any nicotine-containing products. A non-smoker is defined as an individual who has abstained from smoking for at least 1 year prior to screening

Exclusion Criteria:

* A positive pre-study Hepatitis B surface antigen or positive Hepatitis C antibody result within 3 months of screening
* Current or chronic history of liver disease, or known hepatic or biliary abnormalities (with the exception of Gilbert's syndrome or asymptomatic gallstones)
* A positive pre-study drug/alcohol screen
* A positive test for HIV antibody
* History of sensitivity to any of the study medications, Intron A or other recombinant interferons, or components thereof or a history of drug or other allergy that, in the opinion of the investigator or GSK Medical Monitor, contraindicates their participation
* History of regular alcohol consumption within 6 months of the study defined as an average weekly intake of >21 units for males or >14 units for females. One unit is equivalent to 8 g of alcohol and the following can be used as a guide: a half-pint (~240 ml) of beer, 1 glass (125 ml) of wine or 1 (25 ml) measure of spirits
* The subject has participated in a clinical trial and has received an investigational product within the following time period prior to the first dosing day in the current study: 30 days, 5 half-lives or twice the duration of the biological effect of the investigational product (whichever is longer)
* The subject is unwilling to abstain from alcohol consumption from 48 hr prior to dosing until discharge from the clinic, and for 24 hr prior to all other out-patient clinic visits
* Exposure to more than four new chemical entities within 12 months prior to the first dosing day
* Unable to refrain from the use of prescription or non-prescription drugs, including vitamins, herbal and dietary supplements (including St John's Wort) within 7 days (or 14 days if the drug is a potential enzyme inducer) or 5 half-lives (whichever is longer) prior to the first dose of study medication, unless in the opinion of the Investigator and GSK Medical Monitor the medication will not interfere with the study procedures or compromise subject safety
* History of malignancy, except for adequately treated non-invasive cancer of the skin (basal or squamous cell) or cervical carcinoma in situ (>2 yrs prior to dosing)
* Where participation in the study would result in donation of blood or blood products in excess of 500 mL within a 56 day period
* Subjects with a history of or a current thyroid disease or epilepsy
* Subjects exposed to radiation in the 6 months, (except for X-ray/CT examinations of the extremities) prior to the first GFR assessment (Day -2) (cohort B only)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2012-04-30 (Actual); Primary Completion 2012-07-31 (Actual); Study Completion 2012-07-31 (Actual)

PRIMARY OUTCOMES:
Adverse event reporting | Day 1 through to within 7-10 days after the last dose
  Change in health of subjects
Change from baseline in clinical chemistry, hematology, urinalysis | Cohort A: D-1, predose (each session), D2 (each session) and 7-10 days after the last dose. Cohort B single dose session: D-3, predose, D2. Cohort B repeat dose session: D1, D2, D5, D10, D11, D14 and within 7-10 days after last dose
  Change in clinical chemistry, hematology and urinalysis from baseline
Change from baseline in vital signs parameters | Cohort A: Predose, 2h post dose, D2, within 7-10 days from last dose. Cohort B single dose session: D-3, predose, 2h post-dose, D2. Cohort B repeat dose session: predose on D1, D2, D5, D10, 2h post-dose on D1 and D10, D14, within 7-10 days post last dose
  Change in blood pressure, heart rate and body temperature outside normal range
Change from baseline in ECG parameters | Cohort A: Predose, 2h post dose, D2 and within 7-10 days of last dose. Cohort B single dose session: D-3, pre-dose, 2h post-dose and D2. Cohort B repeat dose session: pre-dose, D2, D5, D10, 2h post-dose on D1, D10, D14 and within 7-10 days from last dose
  Change in ECG parameters outside normal range
Plasma concentrations of GSK2586184 | Cohort A: 0.25, 0.5, 1, 2, 4, 8, 12, 24 and 48h post-dose. Cohort B single dose session:0.25, 0.5, 1, 2, 4, 8, 12, 24 and 48h post-dose. Cohort B repeat dose session: D1 and D10 (predose, 0.25, 0.5, 1, 2, 4, 8 and 12h post-dose), D2, D3, D4, D5, and D11
  Change in plasma concentrations of GSK2586184
Change from baseline for 24h urine albumin, creatinine and PCR | Cohort B repeat dose: D-1, D10 and within 7-10 days post last dose
  Change in 24h urine creatinine, albumin and PCR values outside normal range

SECONDARY OUTCOMES:
mRNA expression of IFNa and JAK pathway genes | Cohort B repeat dose: Predose, 1, 2, 4, 8 and 12h on D1 and D10. Predose, 1, 2, 4, 8, 12 and 24h post-dose on D11
  Change in mRNA expression profile of IFNa and JAK pathway genes
Vital signs as a pharmacodynamic endpoint | Cohort B repeat dose: Predose, 4, 8, 12, 24, 28, 32, 48, 72, 100 and 120h post dose on D11
  Change in blood pressure, heart rate and body temperature post IFNa challenge
Plasma levels of Neopterin and B2-microglobulin | Cohort B repeat dose: Predose, 4, 8, 12, 24, 28, 32, 48, 72, 100 and 120h post dose on D11
  Change in plasma concentrations of neopterin and B2-microglobulin post IFNa challenge
Glomerular Filtration Measurement using Cr-51 EDTA | Cohort B: 2h and 4h post Cr-51 EDTA injection on D-2 of single dose session, D8 of repeat dose session and within 7-10 days post last dose
  Change in plasma concentrations of Cr-51 EDTA and it's derived clearance
Duodenal concentrations of GSK2586184 and its metabolites and derived pharmacokinetic parameters | Cohort A: D-1 to D1 predose and 2.5h post-dose to 6.5h post-dose. Cohort B single dose: D-1 to D1 predose and 2.5h post-dose to 6.5h post-dose
  Change in bile concentrations of GSK2586184 and it's metabolites
Urine concentrations of GSK2586184 and its metabolites and derived pharmacokinetic parameters | Cohort A: D1 predose and for 24 hr post-dose.Cohort B single dose: D1 predose and for 24h post-dose
  Change in urine concentration of GSK2586184 and it's metabolites

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Antwerp, Belgium

REFERENCES:
- See also: Results for study 116439 can be found on the GSK Clinical Study Register. — https://gsk-clinicalstudyregister.com/study/116439?search=study&study_ids=116439#rs